CLINICAL TRIAL: NCT03837756
Title: Combining a TLR9 Agonist With Broadly Neutralizing Antibodies for Reservoir Reduction and Immunological Control of HIV Infection: An Investigator-initiated Randomized, Placebo-controlled, Phase IIa Trial.
Brief Title: Combining TLR9 Agonist With bNAbs for Reservoir Reduction and Immunological Control of HIV
Acronym: TITAN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aalborg University Hospital (Other); Odense University Hospital (Other); Rigshospitalet, Denmark (Other); Hvidovre University Hospital (Other); The Peter Doherty Institute for Infection and Immunity (Other); University of Utah (Other); Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: TITAN-001; 2018-001165-16 (EudraCT Number); AGR-2016-8833 (Other Grant/Funding Number: Gilead Sciences, Inc.)
Record Dates: First submitted 2019-02-07; First posted 2019-02-12 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: HIV-1-infection
MeSH Terms: interventions — Sodium Chloride; MGN1703

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1:1:1 in a blinded fashion to receive:
  Arm A: Placebo and Placebo Arm B: Lefitolimod and Placebo Arm C: Placebo and 3BNC117+10-1074 Arm D: Lefitolimod and 3BNC117+10-1074
Who Masked: Participant, Investigator
Masking Description: The participant and all study personnel who directly interact with study participants are blinded to study arm designation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Arm A: Placebo/Placebo (Placebo Comparator): This arm will receive placebo (sterile saline) for both Lefitolimod and 3BNC117 + 10-1074.
  Interventions: Drug: Saline
- Arm B: Lefitolimod/Placebo (Active Comparator): This arm will receive Lefitolimod and placebo (sterile saline) for 3BNC117 + 10-1074.
  Interventions: Drug: Saline; Drug: Lefitolimod
- Arm C: Placebo/3BNC117 + 10-1074 (Active Comparator): This arm will receive 3BNC117 + 10-1074 and placebo (sterile saline) for Lefitolimod.
  Interventions: Drug: Saline; Drug: 3BNC117 and 10-1074
- Arm D: Lefitolimod/3BNC117 + 10-1074 (Active Comparator): This arm will receive both Lefitolimod and 3BNC117 + 10-1074.
  Interventions: Drug: Lefitolimod; Drug: 3BNC117 and 10-1074

INTERVENTIONS:
Drug: Saline — Placebo
  Arms: Arm A: Placebo/Placebo; Arm B: Lefitolimod/Placebo; Arm C: Placebo/3BNC117 + 10-1074
Drug: Lefitolimod — A TLR9 agonist administered s.c. once weekly for 8 weeks.
  Other Names: MGN1703
  Arms: Arm B: Lefitolimod/Placebo; Arm D: Lefitolimod/3BNC117 + 10-1074
Drug: 3BNC117 and 10-1074 — Broadly neutralizing antibodies against HIV env administered two times with a 3 week interval.
  Other Names: RUhumab-001 and RUhumab-002
  Arms: Arm C: Placebo/3BNC117 + 10-1074; Arm D: Lefitolimod/3BNC117 + 10-1074

SUMMARY:
This study is designed to evaluate the safety and efficacy of lefitolimod and 3BNC117/10-1074 in HIV-1-infected individuals on ART and during ATI as intervention to reduce the HIV-1 reservoir

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV-1 infection
* Adults age 18-65 years
* On ART for a minimum of 18 months.
* CD4+ T cell count >500 at screening
* HIV-1 RNA plasma level of < 50 copies/mL by standard assays for at least 15 months (a single viral load measurement > 50 but < 500 copies/mL during this time period is allowable).
* Able to give informed consent
* Viral reservoir sensitivity to 3BNC117 and 10-1074. (Sensitivity of the viral reservoir to neutralization by 3BNC117 and 10-1074 will be tested following the screening visit (i.e. prior to randomization)).

Sensitivity of the viral reservoir to neutralization by 3BNC117 and 10-1074 will be tested following the screening visit (i.e. prior to enrollment and randomization). Isolated PBMCs will be analyzed using the PhenoSense HIV mAb Assay, Monogram Biosciences. The sensitivity of an individuals archieved proviruses to bNAb neutralization will be determined by the IC50 value of PBMC derived pseudovirus inhibition. Subjects that are considered sensitive to both 3BNC117 (IC90<=1.5 μg/mL) and 10-1074 (IC90<=2.0 μg/mL) AND MPI>97 AND fulfill the other inclusion/exclusion criteria will proceed to study enrolment and randomization.

If sensitivity cannot be determined by the PhenoSense HIVmAb Assay, participants will be screened for 3BNC117 and 10-1074 sensitivity using HIV env sequencing carried out in-house (Aarhus, Denmark). The method was originally established and validated by Rockefeller University that already has this method implemented. The method utilizes HIV-1 DNA envelope sequencing and a mathematical prediction binding algoritm of known binding sites of the antibodies. Based on the individual HIV env sequence, proviruses are categorized as "sensitive" or "resistant". Subjects that are determined to be sensitive to both 3BNC117 and 10-1074 (defined as at least 90% of known sequences sensitive to either bNAb) AND fulfill the other inclusion/exclusion criteria will proceed to study enrolment and randomization.

Exclusion Criteria:

* Any significant acute medical illness requiring hospitalization in the past 4 weeks
* Any evidence of an active AIDS-defining opportunistic infection
* Any condition that, in the Investigator's opinion, will prevent adequate compliance with study therapy
* The following laboratory values at screening, the values can be repeated within the screening period, but test results must be available before baseline (Day 0) and checked for eligibility: Hepatic transaminases (AST or ALT) ≥3 x upper limit of normal (ULN) // Serum total bilirubin ≥3 ULN // Estimated glomerular filtration rate (eGFR) ≤50 mL/min (based on serum creatinine) // Platelet count ≤100 x109/L // Absolute neutrophil count ≤1x109/L
* Hepatitis B or C infection
* History of: Malignancy, excluding non-melanoma skin cancers, or organ transplantation
* Receipt of strong immunosuppressive or systemic chemotherapeutic agents within 28 days prior to study entry
* Known resistance to >2 classes of ART
* Known hypersensitivity to the components of lefitolimod, 3BNC117, 10-1074 or their analogues
* Pre-existing autoimmune or antibody-mediated diseases
* Women who are pregnant or breastfeeding, or unwilling/ unable to use an acceptable method of contraception (if of child bearing potential)
* Males or females who are unwilling or unable to use barrier contraception during sexual intercourse until plasma HIV-1 RNA is undetectable using standard assays

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Time to re-initiation of cART during analytical treatment interruption (ATI) | Up to 26 weeks.
  Time from date of cART cessation to the date of the last of three consecutive plasma HIV-1 RNA measurements >10,000 copies/mL, CD4 cell count <350 on two consecutive measurements, or end of ATI (i.e. 26 weeks after cessation of cART) - whichever comes first.

SECONDARY OUTCOMES:
Safety and Tolerability assessment measured by AEs, Adverse Reactions (ARs), SAEs, | Duration of the study
  Subject who receives at least one dose of the IMP(s) will be included in the evaluation for safety, measured by AEs, Adverse Reactions (ARs), SAEs, Serious ARs (SARs) and (SUSAR)
Plasma HIV RNA doubling time | Duration of ATI (up to 26 weeks)
  Plasma HIV RNA doubling time from first measurement >50 copies/mL to first measurement >1,000 copies/mL during the analytical treatment interruption (plasma HIV RNA measured by standard clinical assays, e.g. Cobas TaqMan; Lower limit of quantitation 20 copies/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Ole S Søgaard, MD PhD, Principal Investigator — Aarhus University Hospital
Locations (8):
- Dept. of Internal Medicine, University of Utah, Salt Lake City, Utah, United States
- Alfred Hospital and Monash University, Melbourne, Australia
- Denmark (5):
  - Dept. of Infectious Diseases, Aalborg University Hospital, Aalborg
  - Dept. of Infectious Diseases, Aarhus University Hospital, Aarhus
  - Dept. of Infectious Diseases, Rigshospitalet, Copenhagen
  - Dept. of Infectious Diseases, Amager and Hvidovre Hospitals, Hvidovre
  - Dept. of Infectious Diseases, Odense University Hospital, Odense
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
Individual deidentified participant data (including data dictionaries) will be shared following the publication of the primary and secondary endpoints as outlined in this protocol. Data to be shared includes deidentified data points in published, peer-reviewed articles. Additional, related documents will also be available (study protocol, informed consent form, statistical analysis plan).
Supporting Information: Study Protocol, ICF
Time Frame: Data will become available following publication of the specific dataset with no planned end date.
Access Criteria: Access to the data sharing will be given to researchers who provide a methodologically sound proposal for any type of analysis and requires IRB/Ethics committee approval (if applicable). Proposal should be addressed to olesoega@rm.dk

REFERENCES:
- [Derived] Gunst JD, Hojen JF, Pahus MH, Rosas-Umbert M, Stiksrud B, McMahon JH, Denton PW, Nielsen H, Johansen IS, Benfield T, Leth S, Gerstoft J, Ostergaard L, Schleimann MH, Olesen R, Stovring H, Vibholm L, Weis N, Dyrhol-Riise AM, Pedersen KBH, Lau JSY, Copertino DC Jr, Linden N, Huynh TT, Ramos V, Jones RB, Lewin SR, Tolstrup M, Rasmussen TA, Nussenzweig MC, Caskey M, Reikvam DH, Sogaard OS. Impact of a TLR9 agonist and broadly neutralizing antibodies on HIV-1 persistence: the randomized phase 2a TITAN trial. Nat Med. 2023 Oct;29(10):2547-2558. doi: 10.1038/s41591-023-02547-6. Epub 2023 Sep 11. PMID 37696935